CLINICAL TRIAL: NCT06185478
Title: Prostate Diffusion Imaging With Distortion Correction
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 250301 (15-02-19)
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging (Experimental)
  Interventions: Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: MRI scan — MRI scan

SUMMARY:
There has been literature demonstrating the effectiveness of correcting these MRI images by using an additional measurement of the magnetic field, but the implied improvement in lesion detection in these common distorted regions in the prostate has yet to be shown.

We propose that introducing this distortion correction would greatly improve the DWI images used for tumour detection. For this study we propose testing this hypothesis as a primary objective, and as a secondary objective including additional b-values to further refine the ADC value. The study involves adding one additional distortion correcting scan to the standard clinical study, adding approximately 2 minutes to the study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18 and over
* No contraindication to MR scanning
* Smokers and non-smokers
* Patients who have had a complete scan on the 3T scan MRI at Norfolk and Norwich University Hospital and have gone on to have a biopsy at the Norfolk and Norwich University Hospital

Exclusion Criteria:

* Previous diagnosis of prostate cancer, prostatic biopsy or treatment for prostate cancer

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
MRI image quality | 12 months
  To determine whether correcting for the distortion in MRI images caused by rectal gas improves the image quality and thus diagnostic ability in localising and detecting prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Paul Malcolm, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom